CLINICAL TRIAL: NCT05719649
Title: The Efficacy of NTU 101 Lactic Acid Bacteria Powder in the Adjuvant Improvement of Atopic Dermatitis - A Double-blind, Multi-center Randomized, Placebo-controlled Clinical Trial
Brief Title: The Efficacy of NTU 101 Lactic Acid Bacteria Powder in the Adjuvant Improvement of Atopic Dermatitis Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SunWay Biotech Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21 NTU 101; N202211025 (Other: Office of Human Research, TMU)
Record Dates: First submitted 2023-01-10; First posted 2023-02-09 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis Eczema
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Test group: NTU 101 Lactobacillus Vegetable Capsules Product ingredients: microcrystalline cellulose, corn starch, NTU 101 lactic acid bacteria powder (1.8 x 10^10 CFU); capsule shell composition: HPMC (hydroxypropyl methylcellulose), pure water, titanium dioxide, gellan gum.
Who Masked: Participant, Care Provider
Masking Description: With the random assignment system of Taipei Medical University, 6 Blocks, double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic NTU 101 Lactic Acid Bacteria Capsules (Experimental): The subjects who meet the conditions of this test are randomly assigned according to the ratio of 1:1, and take the lactic acid bacteria NTU 101 (1.8 x 10 ^10 CFU) or Placebo in the test group for a total of 12 weeks of treatment. Once, after the treatment, the test physician evaluated the safety and efficacy of the subjects taking the test group lactobacillus NTU 101.
  Interventions: Dietary Supplement: Lactic acid bacteria NTU 101
- Placebo Capsules (Placebo Comparator): Maltodextrin was used as a placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactic acid bacteria NTU 101 — One NTU 101 Lactic Acid Bacteria Vegetable Capsule a day for a total of 12 weeks.
  Product ingredients: microcrystalline cellulose, corn starch, NTU 101 Lactobacillus paracasei subsp. paracasei NTU 101 (1.8 x 10^10 CFU); capsule shell composition: HPMC (hydroxypropyl methylcellulose), purified water, titanium dioxide, gellan gum.
  Arms: Probiotic NTU 101 Lactic Acid Bacteria Capsules
Dietary Supplement: Placebo — Maltodextrin was used as a placebo
  Arms: Placebo Capsules

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, parallel-controlled trial (14 weeks in total), divided into three periods (screening, treatment, and discontinuation follow-up)

DETAILED DESCRIPTION:
There is a screening period of about 2 weeks before the start of the test product. The subjects who meet the conditions of this test are randomly assigned according to the ratio of 1:1, and take the lactic acid bacteria NTU 101 or Placebo in the test group for a total of 12 weeks of treatment. Once, after the treatment, the test physician evaluated the safety and efficacy of the subjects taking the test group lactobacillus NTU 101 or Placebo.

After the end of the treatment period, all subjects underwent a 2-week discontinuation follow-up period.

This study will track subjects before and after taking samples, SCORing Atopic Dermatitis (Screen-Visit 4), Children's Dermatology Life Quality Index (Visit 1-Visit4), Patient-Oriented Eczema Measure (Visit 1-Visit4), to evaluate subjects Severity of illness.

The subjects received the following tests before and after taking the samples: a full set of blood tests, leukocyte differential counts, serum biochemical tests (BUN, Creatinine, GOT, GPT), and collection of peripheral blood mononuclear cells and stool samples for analysis of the subjects immune function and gastrointestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

- According to the diagnostic criteria of Hanifin & Rajka atopic dermatitis, patients with clinical diagnosis of atopic dermatitis were screened and those who met the following conditions:

1. Age: Children over 6 years old and under 12 years old
2. Patients with moderate atopic dermatitis: SCORAD index 25 - 49.9 (moderate).
3. Atopic dermatitis diagnosed over 6 months

Exclusion Criteria:

1. Immunodeficiency:

   Congenital immunodeficiency: According to the classification principle of "Current classification and status of primary immunodeficiency diseases in Taiwan", it is divided into (1) cellular/T-cell immunodeficiency (2) humoral immunodeficiency (Humoral/B- (3) Complement deficiency (4) Phagocyte deficiency.
2. Human immunodeficiency virus (Human Immunodeficiency Virus, HIV) infection (Inquired from medical records).
3. Other diseases that affect immune function, including kidney disease, diabetes, liver cirrhosis and chronic liver disease, asplenia.
4. Short Bowel Syndrome (Short Bowel Syndrome).
5. Patients with malignant tumors.
6. Patients with central venous catheters.
7. Secondary bacterial infection.
8. Received immunosuppressive and biological agents in the past 3 months (eg: dupilumab, Janus kinase (JAK) inhibitors, Janus kinase inhibitors).
9. Received oral or injectable steroids, antibiotics, and light therapy in the past 1 month.
10. Continuously (3 days or more) take Chinese herbal medicine, probiotic supplements or other fermented foods, such as yogurt, yogurt, and Yakult.
11. Abnormal liver or kidney function (1.5 times higher than normal).
12. Other skin diseases or other systemic diseases.
13. Participated in other clinical trials in the past 3 months.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-14 (Estimated)

PRIMARY OUTCOMES:
SCORing Atopic Dermatitis (SCORAD) Improvement Total Score | 12 weeks
  Compared with the placebo group, after taking probiotics or placebo for 4, 8, and 12 weeks, the atopic dermatitis severity score SCORAD in the control group improved by at least 30% or the ratio of subjects in the test group to the placebo groupPlacebo group According to the statistical method, there is a statistical difference in the total score of SCORAD improvement, at least reaching one of the two items.

CONTACTS AND LOCATIONS:
Overall Officials: Woan-Ruoh Lee, Ph. D., Principal Investigator — Director of Dermatology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Irvine AD, Mina-Osorio P. Disease trajectories in childhood atopic dermatitis: an update and practitioner's guide. Br J Dermatol. 2019 Nov;181(5):895-906. doi: 10.1111/bjd.17766. Epub 2019 May 15. PMID 30758843
- [Result] Doron S, Snydman DR. Risk and safety of probiotics. Clin Infect Dis. 2015 May 15;60 Suppl 2(Suppl 2):S129-34. doi: 10.1093/cid/civ085. PMID 25922398
- [Result] Zuntar I, Petric Z, Bursac Kovacevic D, Putnik P. Safety of Probiotics: Functional Fruit Beverages and Nutraceuticals. Foods. 2020 Jul 17;9(7):947. doi: 10.3390/foods9070947. PMID 32708933
- [Result] Leung DY, Boguniewicz M, Howell MD, Nomura I, Hamid QA. New insights into atopic dermatitis. J Clin Invest. 2004 Mar;113(5):651-7. doi: 10.1172/JCI21060. PMID 14991059
- [Result] Zheng T, Yu J, Oh MH, Zhu Z. The atopic march: progression from atopic dermatitis to allergic rhinitis and asthma. Allergy Asthma Immunol Res. 2011 Apr;3(2):67-73. doi: 10.4168/aair.2011.3.2.67. Epub 2011 Feb 14. PMID 21461244
- [Result] Kim J, Kim BE, Leung DYM. Pathophysiology of atopic dermatitis: Clinical implications. Allergy Asthma Proc. 2019 Mar 1;40(2):84-92. doi: 10.2500/aap.2019.40.4202. PMID 30819278
- [Result] Thyssen JP, Kezic S. Causes of epidermal filaggrin reduction and their role in the pathogenesis of atopic dermatitis. J Allergy Clin Immunol. 2014 Oct;134(4):792-9. doi: 10.1016/j.jaci.2014.06.014. Epub 2014 Jul 25. PMID 25065719
- [Result] McAleer MA, Irvine AD. The multifunctional role of filaggrin in allergic skin disease. J Allergy Clin Immunol. 2013 Feb;131(2):280-91. doi: 10.1016/j.jaci.2012.12.668. PMID 23374260
- [Result] Tsakok T, Woolf R, Smith CH, Weidinger S, Flohr C. Atopic dermatitis: the skin barrier and beyond. Br J Dermatol. 2019 Mar;180(3):464-474. doi: 10.1111/bjd.16934. Epub 2018 Oct 10. PMID 29969827
- [Result] Egawa G, Kabashima K. Barrier dysfunction in the skin allergy. Allergol Int. 2018 Jan;67(1):3-11. doi: 10.1016/j.alit.2017.10.002. Epub 2017 Nov 16. PMID 29153780
- [Result] Reddel S, Del Chierico F, Quagliariello A, Giancristoforo S, Vernocchi P, Russo A, Fiocchi A, Rossi P, Putignani L, El Hachem M. Gut microbiota profile in children affected by atopic dermatitis and evaluation of intestinal persistence of a probiotic mixture. Sci Rep. 2019 Mar 21;9(1):4996. doi: 10.1038/s41598-019-41149-6. PMID 30899033
- [Result] Wakugawa M, Hayashi K, Nakamura K, Tamaki K. Evaluation of mite allergen-induced Th1 and Th2 cytokine secretion of peripheral blood mononuclear cells from atopic dermatitis patients: association between IL-13 and mite-specific IgE levels. J Dermatol Sci. 2001 Feb;25(2):116-26. doi: 10.1016/s0923-1811(00)00118-3. PMID 11164708
- [Result] Czarnowicki T, Santamaria-Babi LF, Guttman-Yassky E. Circulating CLA+ T cells in atopic dermatitis and their possible role as peripheral biomarkers. Allergy. 2017 Mar;72(3):366-372. doi: 10.1111/all.13080. Epub 2016 Dec 15. PMID 27861978
- [Result] Ferran M, Romeu ER, Rincon C, Sagrista M, Gimenez Arnau AM, Celada A, Pujol RM, Hollo P, Jokai H, Santamaria-Babi LF. Circulating CLA+ T lymphocytes as peripheral cell biomarkers in T-cell-mediated skin diseases. Exp Dermatol. 2013 Jul;22(7):439-42. doi: 10.1111/exd.12154. PMID 23800052
- [Result] Czarnowicki T, Esaki H, Gonzalez J, Malajian D, Shemer A, Noda S, Talasila S, Berry A, Gray J, Becker L, Estrada Y, Xu H, Zheng X, Suarez-Farinas M, Krueger JG, Paller AS, Guttman-Yassky E. Early pediatric atopic dermatitis shows only a cutaneous lymphocyte antigen (CLA)(+) TH2/TH1 cell imbalance, whereas adults acquire CLA(+) TH22/TC22 cell subsets. J Allergy Clin Immunol. 2015 Oct;136(4):941-951.e3. doi: 10.1016/j.jaci.2015.05.049. Epub 2015 Aug 1. PMID 26242300
- [Result] Czarnowicki T, He H, Canter T, Han J, Lefferdink R, Erickson T, Rangel S, Kameyama N, Kim HJ, Pavel AB, Estrada Y, Krueger JG, Paller AS, Guttman-Yassky E. Evolution of pathologic T-cell subsets in patients with atopic dermatitis from infancy to adulthood. J Allergy Clin Immunol. 2020 Jan;145(1):215-228. doi: 10.1016/j.jaci.2019.09.031. Epub 2019 Oct 15. PMID 31626841
- [Result] Galazzo G, van Best N, Bervoets L, Dapaah IO, Savelkoul PH, Hornef MW; GI-MDH consortium; Lau S, Hamelmann E, Penders J. Development of the Microbiota and Associations With Birth Mode, Diet, and Atopic Disorders in a Longitudinal Analysis of Stool Samples, Collected From Infancy Through Early Childhood. Gastroenterology. 2020 May;158(6):1584-1596. doi: 10.1053/j.gastro.2020.01.024. Epub 2020 Jan 18. PMID 31958431
- [Result] Kim JE, Kim HS. Microbiome of the Skin and Gut in Atopic Dermatitis (AD): Understanding the Pathophysiology and Finding Novel Management Strategies. J Clin Med. 2019 Apr 2;8(4):444. doi: 10.3390/jcm8040444. PMID 30987008
- [Result] Vernocchi P, Del Chierico F, Fiocchi AG, El Hachem M, Dallapiccola B, Rossi P, Putignani L. Understanding probiotics' role in allergic children: the clue of gut microbiota profiling. Curr Opin Allergy Clin Immunol. 2015 Oct;15(5):495-503. doi: 10.1097/ACI.0000000000000203. PMID 26258924
- [Result] Fujimura KE, Sitarik AR, Havstad S, Lin DL, Levan S, Fadrosh D, Panzer AR, LaMere B, Rackaityte E, Lukacs NW, Wegienka G, Boushey HA, Ownby DR, Zoratti EM, Levin AM, Johnson CC, Lynch SV. Neonatal gut microbiota associates with childhood multisensitized atopy and T cell differentiation. Nat Med. 2016 Oct;22(10):1187-1191. doi: 10.1038/nm.4176. Epub 2016 Sep 12. PMID 27618652
- [Result] Kim SO, Ah YM, Yu YM, Choi KH, Shin WG, Lee JY. Effects of probiotics for the treatment of atopic dermatitis: a meta-analysis of randomized controlled trials. Ann Allergy Asthma Immunol. 2014 Aug;113(2):217-26. doi: 10.1016/j.anai.2014.05.021. Epub 2014 Jun 20. PMID 24954372
- [Result] Huang R, Ning H, Shen M, Li J, Zhang J, Chen X. Probiotics for the Treatment of Atopic Dermatitis in Children: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Front Cell Infect Microbiol. 2017 Sep 6;7:392. doi: 10.3389/fcimb.2017.00392. eCollection 2017. PMID 28932705
- [Result] Climent E, Martinez-Blanch JF, Llobregat L, Ruzafa-Costas B, Carrion-Gutierrez MA, Ramirez-Bosca A, Prieto-Merino D, Genoves S, Codoner FM, Ramon D, Chenoll E, Navarro-Lopez V. Changes in Gut Microbiota Correlates with Response to Treatment with Probiotics in Patients with Atopic Dermatitis. A Post Hoc Analysis of a Clinical Trial. Microorganisms. 2021 Apr 15;9(4):854. doi: 10.3390/microorganisms9040854. PMID 33921166
- [Result] Rather IA, Bajpai VK, Kumar S, Lim J, Paek WK, Park YH. Probiotics and Atopic Dermatitis: An Overview. Front Microbiol. 2016 Apr 12;7:507. doi: 10.3389/fmicb.2016.00507. eCollection 2016. PMID 27148196
- [Result] Gerasimov SV, Vasjuta VV, Myhovych OO, Bondarchuk LI. Probiotic supplement reduces atopic dermatitis in preschool children: a randomized, double-blind, placebo-controlled, clinical trial. Am J Clin Dermatol. 2010;11(5):351-61. doi: 10.2165/11531420-000000000-00000. PMID 20642296
- [Result] Navarro-Lopez V, Ramirez-Bosca A, Ramon-Vidal D, Ruzafa-Costas B, Genoves-Martinez S, Chenoll-Cuadros E, Carrion-Gutierrez M, Horga de la Parte J, Prieto-Merino D, Codoner-Cortes FM. Effect of Oral Administration of a Mixture of Probiotic Strains on SCORAD Index and Use of Topical Steroids in Young Patients With Moderate Atopic Dermatitis: A Randomized Clinical Trial. JAMA Dermatol. 2018 Jan 1;154(1):37-43. doi: 10.1001/jamadermatol.2017.3647. PMID 29117309
- [Result] Ronnstad ATM, Halling-Overgaard AS, Hamann CR, Skov L, Egeberg A, Thyssen JP. Association of atopic dermatitis with depression, anxiety, and suicidal ideation in children and adults: A systematic review and meta-analysis. J Am Acad Dermatol. 2018 Sep;79(3):448-456.e30. doi: 10.1016/j.jaad.2018.03.017. PMID 30119868
- [Result] Feldman SR, Cox LS, Strowd LC, Gerber RA, Faulkner S, Sierka D, Smith TW, Cappelleri JC, Levenberg ME. The Challenge of Managing Atopic Dermatitis in the United States. Am Health Drug Benefits. 2019 Apr;12(2):83-93. PMID 31057694
- [Result] Drucker AM, Eyerich K, de Bruin-Weller MS, Thyssen JP, Spuls PI, Irvine AD, Girolomoni G, Dhar S, Flohr C, Murrell DF, Paller AS, Guttman-Yassky E. Use of systemic corticosteroids for atopic dermatitis: International Eczema Council consensus statement. Br J Dermatol. 2018 Mar;178(3):768-775. doi: 10.1111/bjd.15928. Epub 2018 Jan 28. PMID 28865094
- [Result] Chan TC, Wu NL, Wong LS, Cho YT, Yang CY, Yu Y, Lai PJ, Chang YT, Shih IH, Lee CH, Chu CY. Taiwanese Dermatological Association consensus for the management of atopic dermatitis: A 2020 update. J Formos Med Assoc. 2021 Jan;120(1 Pt 2):429-442. doi: 10.1016/j.jfma.2020.06.008. Epub 2020 Jun 19. PMID 32564976
- [Result] Bin L, Leung DY. Genetic and epigenetic studies of atopic dermatitis. Allergy Asthma Clin Immunol. 2016 Oct 19;12:52. doi: 10.1186/s13223-016-0158-5. eCollection 2016. PMID 27777593